CLINICAL TRIAL: NCT04261218
Title: A Trial to Assess the Safety, Pharmacodynamic Effects, Pharmacokinetics and Efficacy of the MNK Inhibitor Tomivosertib (eFT508) in Combination With Paclitaxel, Following a Run-in Period of Tomivosertib Monotherapy, in Patients With Advanced Breast Cancer
Brief Title: Safety, Pharmacodynamics, Pharmacokinetics, and Efficacy of Tomivosertib Combined With Paclitaxel in Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Translational Research in Oncology (Other)
Collaborators: Effector Therapeutics (Industry); Stand Up To Cancer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TRIO036
Record Dates: First submitted 2020-01-30; First posted 2020-02-07 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tomivosertib; Paclitaxel

STUDY DESIGN:
Intervention Model Description: All patients will be initially treated with tomivosertib monotherapy for 14 ± 2 days (the run-in period). Once the on-treatment samples for pharmacodynamic (PD) assessments are obtained, weekly paclitaxel will be added to the treatment regimen.
  The first 3 to 9 patients will be part of Group 1. The first 3 patients enrolled in this group will receive tomivosertib at a dose of 100 mg orally twice daily (BID), in fasting conditions, and will be assessed for dose-limiting toxicities (DLTs) during the first cycle of tomivosertib in combination with paclitaxel. Depending on the occurrence/absence of DLTs, this first group of 3 patients may need to be expanded (up to 9 patients) or the trial may proceed to start enrollment in Group 2. Group 2 patients will receive tomivosertib at a dose of 100 mg orally BID during the 'run-in' period, as well as weekly paclitaxel in combination with tomivosertib during the 'post run-in' period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 - Dose Finding (Experimental): The first 3 patients enrolled in Group 1 will receive tomivosertib at a dose of 100 mg orally twice daily (BID), under fasting conditions, and will be assessed for dose limiting toxicities (DLTs) during this 'run-in' period. They will also receive the first cycle of tomivosertib IN COMBINATION with weekly paclitaxel in the 'post run-in' period. Depending on the occurrence/absence of DLTs, this first group of 3 patients may need to be expanded (up to 9 patients) or the trial may proceed to start enrollment in Group 2 (detailed in the arm below).
  Interventions: Drug: tomivosertib; Drug: paclitaxel
- Group 2 - Dose Expansion (Experimental): It is anticipated that Group 2 patients will receive tomivosertib at a dose of 100 mg orally twice daily (BID) during the 'run-in' period, which is taken in combination with weekly paclitaxel (according to market label) during the 'post run-in' period.
  Interventions: Drug: tomivosertib; Drug: paclitaxel

INTERVENTIONS:
Drug: tomivosertib — Tomivoserib is supplied as a 100 mg capsule, to be taken orally.
  Other Names: eFT508
Drug: paclitaxel — Taken weekly according to the current market label in combination with experimental tomivosertib.

SUMMARY:
This is a multicenter, open-label trial to evaluate the safety, pharmacodynamics (PD), pharmacokinetics (PK), and efficacy of tomivosertib in combination with paclitaxel in patients with advanced breast cancer (ABC) of any subtype.

The trial will enroll up to 45 patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2 with any breast cancer (BC) subtype and at least one measurable lesion, for whom standard-of-care treatments are ineffective, not tolerated or were refused.

All patients will be initially treated with tomivosertib for 14 days (referred as the run-in period). Once treatment samples are obtained, weekly paclitaxel will be added to the treatment regimen.

Tumor assessments will be done at screening and then periodically throughout trial treatment. Patients will continue to receive trial treatment until progressive disease, as defined according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, intolerable trial-treatment-related toxicity, consent withdrawal, or other criteria is met (defined within the trial protocol).

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Patient Informed Consent Form (PICF) obtained prior to any trial-specific screening procedure.
2. Women or men aged ≥ 18 years-old on the day of the written informed consent is given.
3. Histologically or cytologically confirmed breast adenocarcinoma that is either metastatic (stage IV of the TNM classification) or locally recurrent and not amenable to local curative treatment.
4. Known ER, PgR and HER2 statuses (note: the BC subtype at trial entry will be determined by the statuses in the most recent sample(s) tested for ER, PgR and HER2).
5. Evidence of measurable disease (according to RECIST v.1.1) based on imaging studies and/or physical examination.
6. Patient is a candidate for weekly paclitaxel as palliative treatment for the locally recurrent and/or metastatic disease in the opinion of the treating physician, or is currently receiving paclitaxel (achieving disease control or not). Note: any number of prior lines of standard-of-care or experimental therapies are allowed.
7. At least one metastatic (or recurrent) lesion that is amenable to repeated biopsy and willingness and ability to undergo two biopsies (at screening and approximately 2 weeks after the start of trial treatment).
8. ECOG performance status of 0, 1 or 2.
9. Life expectancy of ≥ 6 months per Investigator's judgement.
10. Adequate organ function during screening, as defined below:

    * Hemoglobin ≥8.0 g/dL (criterion must be met without erythropoietin dependency and without packed red blood cell transfusion within the last 2 weeks)
    * Absolute neutrophil count ≥1,500 cells/mm3
    * Platelet count ≥100,000 cells/mm3
    * Total bilirubin ≤1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
    * Aspartate aminotransferase and alanine aminotransferase ≤3 × ULN (≤5 × ULN for patients with liver metastases)
    * Measured or calculated creatinine clearance (CrCl) >60 mL/min (if calculated, it should be done using the Cockcroft-Gault formula)
11. For women of childbearing potential (WoCBP) - must meet all of the following criteria:

    * Not pregnant (negative serum pregnancy within 14 days of enrollment), and
    * Not breastfeeding, and
    * Willing to use a protocol-recommended method of contraception (refer to details within protocol), from the start of tomivosertib until at least 30 days after the last dose of trial treatment.

    Note: A female patient is considered to be of childbearing potential unless she has had a hysterectomy, bilateral tubal ligation/occlusion, or bilateral oophorectomy, has medically documented ovarian failure (with serum estradiol and follicle-stimulating hormone levels within the institutional laboratory postmenopausal range), or is postmenopausal. Post-menopausal status is defined as 12 consecutive months with no menses without an alternative medical cause.
12. For sexually active male subjects who can father a child - must be willing to refrain from sperm donation and to use a protocol-recommended method of contraception (detailed within protocol), from the start of tomivosertib until at least 74 days after the last dose of trial treatment.
13. Willing and able to comply with the scheduled visits, drug administration plan, protocol-specified laboratory tests, other trial procedures, and trial restrictions. Note: psychological, social, familial, or geographical factors that might preclude adequate trial participation should be considered.

Exclusion Criteria:

1. Current evidence of incomplete recovery from clinically-significant toxicities associated with prior anti-cancer treatment(s), that would represent a contra-indication to experimental therapy in the opinion of the Investigator.
2. Prior systemic standard or investigational anti-cancer therapy within 3 weeks prior to enrollment and/or major surgery within 2 weeks prior to enrollment.
3. Known symptomatic brain metastases requiring ≥10 mg/day of prednisolone (or its equivalent). Patients with previously diagnosed brain metastases are eligible if they have completed their treatment, have recovered from the acute effects of radiation therapy or surgery prior to the start of tomivosertib, fulfill the steroid requirement and are neurologically stable.
4. Active infection requiring systemic therapy.
5. Gastrointestinal disease that may interfere with drug absorption or with interpretation of gastrointestinal adverse events (e.g., gastric or intestinal bypass surgery, pancreatic enzyme insufficiency, malabsorption syndrome, symptomatic inflammatory bowel disease, chronic diarrheal illness, bowel obstruction).
6. Significant cardiovascular disease including myocardial infarction, arterial thromboembolism, or cerebrovascular thromboembolism, within 8 weeks prior to the start of tomivosertib; unstable dysrhythmias or other known clinically significant electrocardiogram abnormality; unstable angina; New York Heart Association Class 3 or 4 congestive heart failure; uncontrolled hypertension (diastolic blood pressure ≥100 mmHg and/or systolic blood pressure ≥180 mmHg); or history of congenital prolonged QT syndrome.
7. Prior therapy with any inhibitor of MNK1 and/or MNK2.
8. Have used a strong inhibitor or inducer of cytochrome P450 (CYP) 3A4, CYP2C9, CYP2D6, or CYP1A2 within 7 days prior to randomization or are expected to require use of a strong inhibitor or inducer of CYP3A4, CYP2C9, CYP2D6, or CYP1A2 during study participation.
9. Known or suspected hypersensitivity to the trial drugs or excipients contained in the trial drugs.
10. History of another malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin; in situ cervical carcinoma; adequately treated, papillary, noninvasive bladder cancer; other adequately treated malignancy currently in complete remission for ≥2 years.
11. History or current evidence of any other medical or psychiatric condition or addictive disorder, or laboratory abnormality that, in the opinion of the Investigator, will increase the risks associated with trial participation, or require treatments that will interfere with the conduct of the trial or the interpretation of trial results.
12. Pregnant or breast-feeding (lactating) women or women who plan to become pregnant or breast-feed during her trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-07-04 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Adverse Events (AEs) | Every serious adverse event (SAE) and related AE, following informed consent and at least until the '30-day safety follow-up' visit, will be assessed. All AEs during treatment will also be included.
  The assessment of safety will be based mainly on the frequency of non-serious and serious AEs. The Medical Dictionary for Regulatory Activities will be used to code all AEs to a system organ class and a preferred term. Incidence of AEs will be tabulated by system organ class, preferred term and toxicity grade. Each of these outputs will include for each AE, system organ class and preferred term as reported by the Investigator based on Common Terminology Criteria for Adverse Events (NCI CTCAE). Detailed listings for all adverse events will also be provided.
Change from Baseline Pharmacodynamic Effects (PD) Following 14 Days of Tomivosertib Monotherapy | All enrolled patients will undergo the sampling for PD assessments during screening and after 14 days (± 2 days) of tomivosertib monotherapy.
  The PD evaluations to be performed will include endpoints related to both direct anti-neoplastic and immunomodulatory actions of the drug. A patient will be considered to have a response if one or more of the PD endpoints (listed in the lab manual) differ between baseline and on-study. The PD response rate will be calculated as the percentage of the patients in the PD Population for whom a PD response is observed.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Tumor assessments used to determine ORR will be conducted at screening and every 8 ± 2 weeks from the enrollment date for 12 months, then every 12 ± 2 weeks, until progressive disease, consent withdrawal, or death.
  ORR is defined as the proportion of patients who have a complete response or partial response according to RECIST v.1.1, based on the Investigator's assessment.
Clinical Benefit Rate (CBR) | Tumor assessments used to determine CBR will be conducted at screening and every 8 ± 2 weeks from the enrollment date for 12 months, then every 12 ± 2 weeks, until progressive disease, consent withdrawal, or death.
  CBR is defined as the proportion of patients who have a complete response or partial response or stable disease according to RECIST v.1.1, based on the Investigator's assessment.
Pharmacokinetic Effects (PK) | All patients from Group 1 and 5-8 patients from Group 2 will be considered as the PK subset. Plasma samples will be obtained at the pre-determined time points during cycle 2 - days 1 and 2. Following cycle 1, treatment cycles are 28 days.
  Plasma concentrations of tomivosertib and paclitaxel will be determined using validated liquid chromatography tandem-mass spectrometry assays. Plasma concentrations will be summarized by scheduled time point with descriptive statistics, which will include the n, mean, standard deviation, coefficient of variation (%), median, minimum, and maximum.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pollak, MD, Study Chair — McGill University
Locations (3):
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Vancouver, Vancouver, British Columbia
  - Jewish General Hospital, Montreal, Quebec